CLINICAL TRIAL: NCT06057987
Title: Polish Registry of Coronary Artery Aneurysms and Ectasias. Coronary ARtery Ectasia Database - Poland (CARED-POL).
Brief Title: Coronary Artery Ectasia Database - Poland
Acronym: CARED-POL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Sylwia Iwanczyk, Principal Investigator, Poznan University of Medical Sciences
Other Study IDs: 687/23
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Aneurysm; Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to comprehensively investigate the current prevalence, morphological characteristics, risk factors for the development, complications as well as long-term prognosis of coronary artery aneurysm and ectasia (CAAE) in the Polish population.

Data obtained from the CARED-POL Registry will enable the selection of morphological risk factors for the unfavorable course of CAAE, including the progression and development of giant aneurysms, aneurysm clotting with vessel occlusion, and thromboembolic complications. Comparing the safety and effectiveness of available CAAE treatment methods in individual patient subgroups will allow individualization of treatment, including anticoagulant therapy.

DETAILED DESCRIPTION:
Coronary artery aneurysm or ectasia (CAAE) is a rare vascular pathology diagnosed in 0.15-5.3% of patients undergoing coronary angiography. CAAEs are often diagnosed incidentally, while symptomatic patients experience various complications, including unstable angina, acute myocardial infarction, arrhythmias, or sudden cardiac death. The most common etiology of CAAE is atherosclerosis, Kawasaki disease, or other vasculitis. Detailed pathomechanisms and risk factors of unfavorable courses of CAAE have not yet been known. In addition, the data on Polish patients are limited to case reports, case series, and small groups from major academic centers.

CARED-POL is a multicenter, observational nationwide registry of CAAE. Patients will be included ambispectively based on the angiographic diagnosis of coronary artery aneurysm (CAA) or coronary artery ectasia (CAE).

All participating centers will enroll patients retrospectively based on their internal databases after evaluation of coronary angiography by an experienced interventional cardiologist and prospectively for six months from the CARED-POL joining. Angiographic assessment will be based on quantitative coronary angiography (QCA). The patient data will be collected from standardized and anonymous forms via the Scientific Platform of the Polish Society of Cardiology. In accordance with initial assumptions, 2,000 patients in all participating centers will be included.

Patients included in the registry will undergo a minimum of 6 months of follow-up with assessment of the following endpoints: all-cause death, re-hospitalization for unstable angina, myocardial infarction, heart failure, bleeding, stroke, embolic events, and any cause for repeat coronary angiography.

Data will be obtained from outpatient visits, medical records, or telephone interviews. In patients who undergo repeated coronary angiography, the formation of a new aneurysm or progression of an existing one will be detected. Aneurysm progression is diagnosed as an increase in size demonstrated on at least two orthogonal angiographic views.

ELIGIBILITY:
Inclusion Criteria:

* CAA or CAE defined as a focal dilatation with a diameter of more than or equal to 1.5 times the adjacent normal coronary segment

Exclusion Criteria:

* the lack of informed consent for prospectively enrolled patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included ambispectively based on the angiographic diagnosis of CAA or CAE. CAA is defined as a focal dilatation with a diameter of more than or equal to 1.5 times the adjacent normal coronary segment, while CAE is analogous lesions but more diffuse, exceeding more than a third of the coronary artery length. A giant CAAE is diagnosed when the diameter of the artery exceeded 4-fold the diameter of the reference vessel.
  Each participating center with the cath lab will enroll patients retrospectively from their internal databases after evaluation of coronary angiography by an experienced interventional cardiologist using quantitative coronary angiography (QCA), but also prospectively for 6 months from the CARED-POL joining. The patient data will be collected from standardized and anonymous forms via Scientific Platform of the Polish Society of Cardiology. In accordance with initial assumptions 2,000 patients in all participating centers will be included.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of CAAE | 12 months
  Incidence of CAAE in the Polish population based on coronary angiography
All-cause death | 6 months
Re-hospitalization | 6 months
  Re-hospitalization for unstable angina, myocardial infarction, heart failure, bleeding, stroke, embolic events

CONTACTS AND LOCATIONS:
Overall Officials: Sylwia Iwańczyk, MD, PhD, Principal Investigator — Poznań University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poland, Poznan, Wielkopolska, Poland